CLINICAL TRIAL: NCT03386721
Title: An Open-Label, Multicenter, Phase II Study to Evaluate the Therapeutic Activity of Simlukafusp Alfa (RO6874281), an Immunocytokine, Consisting of Interleukin-2 Variant (IL-2v) Targeting Fibroblast Activation Protein-Α (FAP), in Combination With Atezolizumab (Anti-PD-L1), Administered Intravenously, in Participants With Advanced and/or Metastatic Solid Tumors
Brief Title: Basket Study to Evaluate the Therapeutic Activity of Simlukafusp Alfa as a Combination Therapy in Participants With Advanced and/or Metastatic Solid Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The Sponsor discontinued the development of Simlukafusp alfa due to portfolio prioritization, not due to any safety, efficacy, or quality issues.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BP40234; 2017-003182-94 (EudraCT Number)
Record Dates: First submitted 2017-12-22; First posted 2017-12-29 (Actual); Results first posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Advanced/Metastatic Head and Neck, Oesophageal and Cervical Cancers
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — atezolizumab; Gemcitabine; Vinorelbine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (17):
- Cohort A (Part I) (Experimental): Checkpoint Inhibitor (CPI)-Naïve Participants with non-small-cell lung cancer (NSCLC) who have not received CPI therapy previously will receive simlukafusp alfa intravenous (IV) infusion once in a week (QW) for first 5 doses, and once in 2 weeks (Q2W) for remaining doses up to maximum 36 months. Simlukafusp alfa will be administered at a 10 mg flat dose. Atezolizumab IV infusion will be administered in combination Q2W at a dose of 840 mg. Tumor biopsies: collection of fresh tumor biopsies (at baseline and on-treatment) will be optional.
  Interventions: Drug: simlukafusp alfa; Drug: Atezolizumab (MPDL3280A), an Engineered Anti-PD-L1 Antibody
- Cohort B (Part I) (Experimental): CPI-Experienced Participants (NSCLC) who have received CPI therapy previously will receive simlukafusp alfa intravenous (IV) infusion once in a week (QW) for first 5 doses, and once in 2 weeks (Q2W) for remaining doses up to maximum 36 months. Simlukafusp alfa will be administered at a 10 mg flat dose. Atezolizumab IV infusion will be administered in combination Q2W at a dose of 840 mg. Tumor biopsies: 2 mandatory fresh tumor biopsies, one at baseline and one on-treatment, will be collected. Additional on-treatment biopsies will be optional.
  Interventions: Drug: simlukafusp alfa; Drug: Atezolizumab (MPDL3280A), an Engineered Anti-PD-L1 Antibody
- Cohort C (Part I) (Experimental): This is a mandatory biopsy cohort based on the treatment's safety and preliminary activity analysis to enroll CPI-Naive Participants. Participants (NSCLC) will receive simlukafusp alfa intravenous (IV) infusion once in a week (QW) for first 5 doses, and once in 2 weeks (Q2W) for remaining doses up to maximum 36 months. Simlukafusp alfa will be administered at a 10 mg flat dose. Atezolizumab IV infusion will be administered in combination Q2W at a dose of 840 mg.
  Tumor biopsies: 2 mandatory fresh tumor biopsies, one at baseline and one on-treatment, will be collected. Additional on-treatment biopsies will be optional.
  Interventions: Drug: simlukafusp alfa; Drug: Atezolizumab (MPDL3280A), an Engineered Anti-PD-L1 Antibody
- Cohort D Arm I (Part I) (Experimental): CPI Experienced Participants (NSCLC) who were previously treated with platinum and docetaxel.
  Participants will receive simlukafusp alfa intravenous (IV) infusion once in a week (QW) for first 5 doses, and once in 2 weeks (Q2W) for remaining doses up to maximum 36 months. Simlukafusp alfa will be administered at a 10 mg flat dose. Atezolizumab IV infusion will be administered in combination Q2W at a dose of 840 mg.
  Tumor biopsies: 2 mandatory fresh tumor biopsies, one at baseline and one on-treatment, will be collected. Additional on-treatment biopsies will be optional.
  Interventions: Drug: simlukafusp alfa; Drug: Atezolizumab (MPDL3280A), an Engineered Anti-PD-L1 Antibody
- Cohort D Arm 2 (Part I) (Experimental): CPI Experienced Participants (NSCLC) who were previously treated with platinum and docetaxel.
  Participants will receive simlukafusp alfa intravenous (IV) infusion once in 3 weeks (Q3W) up to maximum 36 months. Simlukafusp alfa will be administered at a 10 mg flat dose. Atezolizumab IV infusion will be administered in combination Q3W at a dose of 1200 mg.
  Tumor biopsies: 2 mandatory fresh tumor biopsies, one at baseline and one on-treatment, will be collected. Additional on-treatment biopsies will be optional.
  Interventions: Drug: simlukafusp alfa; Drug: Atezolizumab (MPDL3280A), an Engineered Anti-PD-L1 Antibody
- Cohort D Arm 3 (Part I) (Experimental): CPI Experienced Participants (NSCLC) who were previously treated with platinum and docetaxel will receive a single-agent gemcitabine or vinorelbine as per approved protocol.
  Tumor biopsies: 2 mandatory fresh tumor biopsies, one at baseline and one on-treatment, will be collected. Additional on-treatment biopsies will be optional.
  Interventions: Drug: Gemcitabine; Drug: Vinorelbine
- Cohort E Arm I (Part II) (Experimental): This cohort will enroll participants (NSCLC) with High-Tumor PD-L1 Expression who have not received any prior systemic therapy. Participants will receive simlukafusp alfa intravenous (IV) infusion once in a week (QW) for first 5 doses, and once in 2 weeks (Q2W) for remaining doses up to maximum 36 months. Simlukafusp alfa will be administered at a 10 mg flat dose. Atezolizumab IV infusion will be administered in combination Q2W at a dose of 840 mg.
  Tumor biopsies: 2 mandatory fresh tumor biopsies, one at baseline and one on-treatment, will be collected. Additional on-treatment biopsies will be optional.
  Interventions: Drug: simlukafusp alfa; Drug: Atezolizumab (MPDL3280A), an Engineered Anti-PD-L1 Antibody
- Cohort E Arm 2 (Part II) (Experimental): This cohort will enroll participants (NSCLC) with High-Tumor PD-L1 Expression who have not received any prior systemic therapy. Participants will receive simlukafusp alfa IV infusion in combination with atezolizumab Q3W. Simlukafusp alfa will be administered at a 10 mg flat dose. Atezolizumab IV infusion will be administered at a dose of 1200 mg.
  Tumor biopsies: 2 mandatory fresh tumor biopsies, one at baseline and one on-treatment, will be collected. Additional on-treatment biopsies will be optional.
  Interventions: Drug: simlukafusp alfa; Drug: Atezolizumab (MPDL3280A), an Engineered Anti-PD-L1 Antibody
- Cohort F (Part I) (Experimental): CPI-experienced, docetaxel naive participants (NSCLC) who experienced disease progression during or following treatment with a platinum - containing regimen. Participants will receive combination of simlukafusp alfa and atezolizumab in a Q3W schedule. Simlukafusp alfa will be administered at a 10 mg flat dose. Atezolizumab IV infusion will be administered at a dose of 1200 mg.
  Tumor biopsies: one mandatory fresh tumor biopsy will be collected at baseline. Additional on-treatment biopsies will be optional.
  Interventions: Drug: simlukafusp alfa; Drug: Atezolizumab (MPDL3280A), an Engineered Anti-PD-L1 Antibody
- Cohort G (Part III) (Experimental): CPI-naïve SCC of the head and neck (SCCHN) (20 response-evaluable participants), mandatory biopsies. Participants in cohort G Part III will receive simlukafusp alfa Q3W in combination with atezolizumab Q3W. Simlukafusp alfa will be administered at a 10 mg flat dose. Atezolizumab IV infusion will be administered at a dose of 1200 mg. Tumor biopsies: one mandatory fresh tumor biopsy will be collected at baseline. Additional on-treatment biopsies will be optional. Biopsies are not applicable to participants presenting with a single target lesion and absence of any non-target lesion.
  Interventions: Drug: simlukafusp alfa; Drug: Atezolizumab (MPDL3280A), an Engineered Anti-PD-L1 Antibody
- Cohort H (Part III) (Experimental): Previously treated, CPI-experienced squamous cell carcinoma head and heck cancer (20 response evaluable participants), mandatory biopsies. Participants in cohort H Part III will receive simlukafusp alfa Q3W in combination with atezolizumab Q3W. Simlukafusp alfa will be administered at a 10 mg flat dose. Atezolizumab IV infusion will be administered at a dose of 1200 mg. Tumor biopsies: one mandatory fresh tumor biopsy will be collected at baseline. Additional on-treatment biopsies will be optional. Biopsies are not applicable to participants presenting with a single target lesion and absence of any non-target lesion.
  Interventions: Drug: simlukafusp alfa; Drug: Atezolizumab (MPDL3280A), an Engineered Anti-PD-L1 Antibody
- Cohort I (Part III) (Experimental): Previously treated, CPI-naïve squamous esophageal cancer (20 response evaluable participants), mandatory biopsies. Participants in cohort I Part III will receive simlukafusp alfa Q3W in combination with atezolizumab Q3W. Simlukafusp alfa will be administered at a 10 mg flat dose. Atezolizumab IV infusion will be administered at a dose of 1200 mg. Tumor biopsies: one mandatory fresh tumor biopsy will be collected at baseline. Additional on-treatment biopsies will be optional.
  Interventions: Drug: simlukafusp alfa; Drug: Atezolizumab (MPDL3280A), an Engineered Anti-PD-L1 Antibody
- Cohort J (Part III) (Experimental): Previously treated, CPI-naïve squamous cervical cancer (20 response evaluable participants): mandatory biopsy. Participants in cohort J Part III will receive simlukafusp alfa Q3W in combination with atezolizumab Q3W. Simlukafusp alfa will be administered at a 10 mg flat dose. Atezolizumab IV infusion will be administered at a dose of 1200 mg. Tumor biopsies: one mandatory fresh tumor biopsy will be collected at baseline. Additional on-treatment biopsies will be optional.
  Interventions: Drug: simlukafusp alfa; Drug: Atezolizumab (MPDL3280A), an Engineered Anti-PD-L1 Antibody
- Cohort K (Part III) (Experimental): CPI-naïve SCC of the head and neck (SCCHN) (20 response-evaluable participants), mandatory biopsies. Participants in cohort K Part III will receive simlukafusp alfa QW in combination with atezolizumab Q2W for 4 weeks followed by simlukafusp alfa in combination with atezolizumab Q2W. Simlukafusp alfa will be administered at a 10 mg flat dose. Atezolizumab IV infusion will be administered at a dose of 840 mg. Tumor biopsies: one mandatory fresh tumor biopsy will be collected at baseline. Additional on-treatment biopsies will be optional. Biopsies are not applicable to participants presenting with a single target lesion and absence of any non-target lesion.
  Interventions: Drug: simlukafusp alfa; Drug: Atezolizumab (MPDL3280A), an Engineered Anti-PD-L1 Antibody
- Cohort L (Part III) (Experimental): Previously treated, CPI-experienced squamous cell carcinoma head and neck cancer (20 response evaluable participants), mandatory biopsies. Participants in cohort L Part III will receive simlukafusp alfa QW in combination with atezolizumab Q2W for 4 weeks followed by simlukafusp alfa in combination with atezolizumab Q2W. Simlukafusp alfa will be administered at a 10 mg flat dose. Atezolizumab IV infusion will be administered at a dose of 840 mg. Tumor biopsies: one mandatory fresh tumor biopsy will be collected at baseline. Additional on-treatment biopsies will be optional. Biopsies are not applicable to participants presenting with a single target lesion and absence of any non-target lesion.
  Interventions: Drug: simlukafusp alfa; Drug: Atezolizumab (MPDL3280A), an Engineered Anti-PD-L1 Antibody
- Cohort M (Part III) (Experimental): Esophageal SCC participants will receive simlukafusp alfa QW in combination with atezolizumab Q2W for 4 weeks followed by simlukafusp alfa in combination with atezolizumab Q2W. Simlukafusp alfa will be administered at a 10 mg flat dose. Atezolizumab IV infusion will be administered at a dose of 840 mg. Tumor biopsies: one mandatory fresh tumor biopsy will be collected at baseline. Additional on-treatment biopsies will be optional.
  Interventions: Drug: simlukafusp alfa; Drug: Atezolizumab (MPDL3280A), an Engineered Anti-PD-L1 Antibody
- Cohort N (Part III) (Experimental): Cervical SCC participants will receive simlukafusp alfa QW in combination with atezolizumab Q2W for 4 weeks followed by simlukafusp alfa in combination with atezolizumab Q2W. Simlukafusp alfa will be administered at a 10 mg flat dose. Atezolizumab IV infusion will be administered at a dose of 840 mg. Tumor biopsies: one mandatory fresh tumor biopsy will be collected at baseline. Additional on-treatment biopsies will be optional.
  Interventions: Drug: simlukafusp alfa; Drug: Atezolizumab (MPDL3280A), an Engineered Anti-PD-L1 Antibody

INTERVENTIONS:
Drug: simlukafusp alfa — simlukafusp alfa will be administered as per the dosage regimen mentioned in arm descriptions.
  Other Names: RO6874281
  Arms: Cohort A (Part I); Cohort B (Part I); Cohort C (Part I); Cohort D Arm 2 (Part I); Cohort D Arm I (Part I); Cohort E Arm 2 (Part II); Cohort E Arm I (Part II); Cohort F (Part I); Cohort G (Part III); Cohort H (Part III); Cohort I (Part III); Cohort J (Part III); Cohort K (Part III); Cohort L (Part III); Cohort M (Part III); Cohort N (Part III)
Drug: Atezolizumab (MPDL3280A), an Engineered Anti-PD-L1 Antibody — Atezolizumab will be administered as per the dosage regimen mentioned in arm descriptions.
  Arms: Cohort A (Part I); Cohort B (Part I); Cohort C (Part I); Cohort D Arm 2 (Part I); Cohort D Arm I (Part I); Cohort E Arm 2 (Part II); Cohort E Arm I (Part II); Cohort F (Part I); Cohort G (Part III); Cohort H (Part III); Cohort I (Part III); Cohort J (Part III); Cohort K (Part III); Cohort L (Part III); Cohort M (Part III); Cohort N (Part III)
Drug: Gemcitabine — Single-agent treatment administered as per approved protocol.
  Arms: Cohort D Arm 3 (Part I)
Drug: Vinorelbine — Single-agent treatment administered as per approved protocol.
  Arms: Cohort D Arm 3 (Part I)

SUMMARY:
This is an open-label, multicenter, basket trial Phase II study to evaluate the antitumor activity of simlukafusp alfa in combination with atezolizumab in participants with advanced and/or metastatic solid tumors. Currently the focus is on participants with Head and Neck, oesophageal and cervical cancers with confirmed squamous cell carcinoma histology type.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have progressed on at least one previous regimen of anticancer therapy (chemotherapy, mutation targeted therapy, and/or CPI therapy)
* Measurable disease, as defined by RECIST Version 1.1
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1 or Karnofsky Performance Score greater than or equal to (>=) 70
* Life expectancy of >=12 weeks
* Confirmed at least one tumor lesion with location accessible to safely biopsy per clinical judgment of the treating physician.

Biopsies are not applicable to participants in Cohorts G, H, K, and L presenting with a single target lesion and absence of any non-target lesion.

* Consent to provide an archival tumor tissue sample (if available, applicable to all participants)
* Willingness to undergo baseline and on-treatment tumor biopsies for pharmacodynamics (PD) biomarker analysis (biopsies are optional for Cohort A)
* Adequate cardiovascular function as defined in the study protocol
* AEs related to any previous radiotherapy, chemotherapy, or surgical procedure must have resolved to Grade less than or equal to (<=) 1, except alopecia (any grade) and Grade 2 peripheral neuropathy
* Adequate haematological, liver, and renal functions.
* Participants with unilateral pleural effusion (indications other than NSCLC) are eligible if they fulfill both of the following:

  1. NYHA Class 1
  2. Forced expiratory volume 1 (FEV1) and forced vital capacity (FVC) >70% of predicted value; participants with lung metastases should present with DLCO >60% of predicted value.
* Participants with Gilbert's syndrome will be eligible for the study
* Participants must have had confirmed diagnosis of recurrent or metastatic squamous cell carcinoma head and neck, or esophageal cancer or metastatic, persistent or recurrent squamous cervical cancer.

Exclusion Criteria:

* Symptomatic or untreated central nervous system (CNS) metastases
* History of treated asymptomatic CNS metastases as described in the protocol
* Spinal cord compression not definitively treated with surgery and/or radiation or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for >=2 weeks before enrollment
* Leptomeningeal disease
* An active second malignancy
* Penetrating tumor infiltration
* Evidence of significant, uncontrolled concomitant diseases that could affect compliance with the protocol or interpretation of results
* Episode of significant cardiovascular/cerebrovascular acute disease within 6 months before study treatment administration
* History of significant vascular disease (for example, aortic aneurysm, aortic dissection)
* Active or uncontrolled infections
* Human immunodeficiency virus (HIV) or Active Hepatitis A, B, C, D or E infection (HAV/HBV/HCV/HDV/HEV).
* Severe infection within 4 weeks before study treatment administration including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia.
* History of chronic liver disease or evidence of hepatic cirrhosis
* Dementia or altered mental status that would prohibit informed consent
* History of, active or suspicion of autoimmune disease
* History of idiopathic pulmonary fibrosis, pneumonitis (including drug-induced), organizing pneumonia (bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis on screening chest computed tomography (CT) scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted
* Bilateral pleural effusion confirmed by X-ray
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding that give reasonable suspicion of a disease or condition that would contraindicate the use of an investigational drug
* Concurrent therapy with any other investigational drug
* Immunomodulating agents as described in study protocol
* Chronic use of steroids
* Last dose with any cytostatic treatments < 28 days before study treatment administration
* Radiotherapy within the last 4 weeks before start of study treatment administration, with the exception of limited field palliative radiotherapy
* Administration of a live, attenuated vaccine within 4 weeks before Cycle 1 Day 1 or at any time during the study and 5 months after the last dose of atezolizumab
* Major surgery or significant traumatic injury <28 days before study treatment administration (excluding fine needle biopsies) or if wound healing has not completed after surgery or anticipation of the need for major surgery during study treatment
* Known hypersensitivity to any of the components of the simlukafusp alfa drug product or atezolizumab drug product
* Severe dyspnea at rest or requiring supplementary oxygen therapy Locally curative options are available for participant's disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2018-02-19 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (44):
- United States (2):
  - University of California, San Francisco, Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Cancer Treatment Centers of America, Newnan, Georgia
- Belgium (3):
  - UZ Antwerpen, Edegem
  - UZ Gent, Ghent
  - UZ Leuven Gasthuisberg, Leuven
- France (4):
  - Institut Bergonie, Bordeaux
  - Hopital Timone Adultes; Oncologie Medicale Et Usp, Marseille
  - ICM; Medecine B3, Montpellier
  - Gustave Roussy Cancer Campus, Villejuif
- Universitätsklinikum Essen; Innere Klinik (Tumorforschung), Essen, Germany
- Rambam Medical Center; Oncology, Haifa, Israel
- Auckland City Hospital; Clinical Oncology, Auckland, New Zealand
- Poland (2):
  - Uniwersyteckie Centrum Kliniczne; Osrodek Badan Wczesnych Faz, Gda?sk
  - Narodowy Instytut Onkologii im. M. Sklodowskiej-Curie; Oddzial Badan Wczesnych Faz, Warsaw
- Russia (2):
  - N.N.Burdenko Main Military Clinical Hospital; Oncology Dept, Moscow
  - S-Pb clinical scientific practical center of specialized kinds of medical care (oncological), Saint Petersburg
- Singapore (2):
  - National University Hospital; National University Cancer Institute, Singapore (NCIS), Singapore
  - National Cancer Centre; Medical Oncology, Singapore
- South Korea (5):
  - Seoul National University Bundang Hospital, Seongnam-si
  - Severance Hospital, Yonsei University Health System, Seoul
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (8):
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Hospital del Mar; Servicio de Oncologia, Barcelona
  - Hospital Univ Vall d'Hebron; Servicio de Oncologia, Barcelona
  - Clinica Universidad de Navarra Madrid; Servicio de Oncología, Madrid
  - Hospital Ramon y Cajal; Servicio de Oncologia, Madrid
  - START Madrid-FJD, Hospital Fundacion Jimenez Diaz, Madrid
  - START Madrid. Centro Integral Oncologico Clara Campal; CIOCC, Madrid
  - Hospital Clinico Universitario de Valencia; Servicio de Onco-hematologia, Valencia
- Hôpitaux Universit. de Genève Médecine Oncologie; Oncologie, Geneva, Switzerland
- Taiwan (2):
  - National Cheng Kung Uni Hospital; Dept of Hematology and Oncology, Tainan
  - National Taiwan Uni Hospital; Dept of Oncology, Taipei
- Turkey (Türkiye) (6):
  - Adana Baskent University Hospital; Medical Oncology, Adana
  - Akdeniz University Medical Faculty; Medical Oncology Department, Antalya
  - Trakya Universitesi Tip Fakultesi, Medikal Onkoloji Bilim Dali, Balkan Yerleskesi, Edirne
  - Istanbul University Cerrahpa?a-Cerrahpa?a Medical Faculty; Medikal Onkoloji Departmani, Istanbul
  - ?zmir Medical Park; Onkoloji, Izmir
  - Goztepe Prof.Dr. Suleyman Yalcin City Hospital; Clinical Oncology, Kadiköy
- United Kingdom (4):
  - Barts, London
  - University College London Hospital, London
  - Christie Hospital Nhs Trust; Medical Oncology, Manchester
  - Royal Marsden Hospital; Institute of Cancer Research, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] Verlingue L, Italiano A, Prenen H, Guerra Alia EM, Tosi D, Perets R, Lugowska I, Moiseyenko V, Gumus M, Arslan C, Lindsay CR, Deva S, Taus A, Oaknin A, Rottey S, Cicin I, Goksu SS, Smolin A, Rosello-Keranen S, Habigt C, Marbach D, Boetsch C, Dejardin D, Sleiman N, Evers S, Richard M, Ardeshir C, Charo J, Kraxner A, Teichgraber V, Keshelava N, Dziadziuszko R. Phase 2 study of the antitumour activity and safety of simlukafusp alfa (FAP-IL2v) combined with atezolizumab in patients with recurrent and/or metastatic cervical squamous cell carcinoma. EBioMedicine. 2024 Nov;109:105374. doi: 10.1016/j.ebiom.2024.105374. Epub 2024 Oct 11. PMID 39395231
- [Derived] Prenen H, Deva S, Keam B, Lindsay CR, Lugowska I, Yang JC, Longo F, de Miguel M, Ponz-Sarvise M, Ahn MJ, Gumus M, Champiat S, Italiano A, Salas S, Perets R, Arslan C, Cho BC, Evers S, Boetsch C, Marbach D, Dejardin D, Sleiman N, Ardeshir C, Richard M, Charo J, Kraxner A, Keshelava N, Teichgraber V, Moreno V. Phase II Study to Determine the Antitumor Activity and Safety of Simlukafusp Alfa (FAP-IL2v) Combined with Atezolizumab in Esophageal Cancer. Clin Cancer Res. 2024 Jul 15;30(14):2945-2953. doi: 10.1158/1078-0432.CCR-23-2677. PMID 38709220

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 42 investigative sites in Belgium, France, Germany, Israel, Korea, New Zealand, Poland, Russia, Singapore, Spain, Switzerland, Taiwan, Turkey, United Kingdom, USA from 19 February 2018 to 30 December 2021
Pre-assignment Details: A total of 256 participants were enrolled. 95 participants in non-small cell lung cancer (NCSLC) cohorts [Part I: A, B, D, F & Part II: E] & 161 participants in squamous cell carcinoma (SCC) cohort (78 with head and neck SCC (HNSCC) [Part III: G, H, K], 35 in esophageal SCC (ESCC) [Part 3: I and M], & 48 in cervical SCC (CSCC) [Part 3 J & N] received simlukafusp alfa & atezolizumab. No participants were enrolled in Cohorts C & L as emerging data did not lead to the need to open these cohorts.
Groups:
- NSCLC: Part I Cohort A (QW/Q2W): Checkpoint Inhibitor (CPI)-naïve participants with NSCLC, received simlukafusp alfa, 10 milligrams (mg), intravenous (IV) infusion, once weekly (QW) for the first 4 weeks, and every 2 weeks (Q2W) until disease progression, unacceptable toxicity, or withdrawal of consent, or for a maximum of 38 months. Participants also received atezolizumab, 840 mg, IV infusion, Q2W in combination with simlukafusp alfa until disease progression, unacceptable toxicity, or withdrawal of consent, or for a maximum of 38 months.
- NSCLC: Part I Cohort B (QW/Q2W): CPI-experienced participants with NSCLC, received simlukafusp alfa, 10 mg, IV infusion, QW for the first 4 weeks, and Q2W until disease progression, unacceptable toxicity, or withdrawal of consent, or for a maximum of 15.6 months. Participants also received atezolizumab, 840 mg, IV infusion, Q2W in combination with simlukafusp alfa until disease progression, unacceptable toxicity, or withdrawal of consent, or for a maximum of 15.6 months.
- NSCLC: Part I Cohort D, Arm 1 (QW/Q2W): CPI-experienced participants with NSCLC previously treated with platinum-containing regimen and docetaxel, received simlukafusp alfa, 10 mg, IV infusion, QW for the first 4 weeks, and Q2W until disease progression, unacceptable toxicity, or withdrawal of consent, or for a maximum of 2.7 months. Participants also received atezolizumab, 840 mg, IV infusion, Q2W in combination with simlukafusp alfa until disease progression, unacceptable toxicity, or withdrawal of consent, or for a maximum of 2.7 months.
- NSCLC: Part I Cohort D, Arm 2 (Q3W): CPI-experienced participants with NSCLC previously treated with platinum-containing regimen and docetaxel received simlukafusp alfa, 10 mg, IV infusion once in 3 weeks (Q3W) in combination with atezolizumab, 1200 mg, IV infusion, Q3W until disease progression, unacceptable toxicity, or withdrawal of consent, or for a maximum of 5.4 months.
- NSCLC: Part I Cohort D, Arm 3 (Q3W): CPI-experienced participants with NSCLC who were previously treated with platinum-containing regimen and docetaxel received a gemcitabine, IV infusion as per approved protocol. Participants who had documented radiographic disease progression during or after treatment with gemcitabine received simlukafusp alfa, 10 mg, IV infusion Q3W in combination with atezolizumab, 1200 mg, IV infusion, Q3W until disease progression, unacceptable toxicity, or withdrawal of consent, or for a maximum of 1.3 months.
- NSCLC: Part I Cohort F (Q3W): CPI-experienced, docetaxel naive participants with NSCLC who experienced disease progression during or after treatment with a platinum-containing regimen received, simlukafusp alfa, 10 mg, IV infusion, Q3W in combination with atezolizumab, 1200 mg, IV infusion, Q3W until disease progression, unacceptable toxicity, or withdrawal of consent, or for a maximum of 26 months.
- NSCLC: Part II Cohort E, Arm 1 (QW/Q2W): NSCLC participants without prior treatment for metastatic disease and with high programmed death-ligand 1 (PD-L1) expression levels, received simlukafusp alfa, 10 mg, IV infusion, QW for the first 4 weeks, and Q2W until disease progression, unacceptable toxicity, or withdrawal of consent, or for a maximum of 31.3 months. Participants also received atezolizumab, 840 mg, IV infusion, Q2W in combination with simlukafusp alfa until disease progression, unacceptable toxicity, or withdrawal of consent, or for a maximum of 31.3 months.
- NSCLC: Part II Cohort E, Arm 2 (Q3W): NSCLC participants without prior treatment for metastatic disease and with high PD-L1 expression levels, received simlukafusp alfa, 10 mg, IV infusion Q3W in combination with atezolizumab, 1200 mg, IV infusion, Q3W until disease progression, unacceptable toxicity, or withdrawal of consent, or for a maximum of 18.6 months.
- SCCHN: Part III Cohort G (Q3W): CPI-naïve participants with SCCHN, received simlukafusp alfa, 10 mg, IV infusion, Q3W in combination with atezolizumab, 1200 mg, IV infusion, Q3W until disease progression, unacceptable toxicity, or withdrawal of consent, or for a maximum of 24.6 months.
- SCCHN: Part III Cohort H (Q3W): CPI-experienced participants with SCCHN, received simlukafusp alfa, 10 mg, IV infusion, Q3W in combination with atezolizumab, 1200 mg, IV infusion, Q3W until disease progression, unacceptable toxicity, or withdrawal of consent, or for a maximum of 10.3 months.
- ESCC: Part III Cohort I (Q3W): CPI-naïve participants with ESCC who were previously treated with standard therapy received simlukafusp alfa, 10 mg, IV infusion, Q3W in combination with atezolizumab, 1200 mg, IV infusion, Q3W until disease progression, unacceptable toxicity, or withdrawal of consent, or for a maximum of 30.5 months.
- CSCC: Part III Cohort J (Q3W): CPI-naïve participants with CSCC who were previously treated with standard therapy, received simlukafusp alfa, 10 mg, IV infusion, Q3W in combination with atezolizumab, 1200 mg, IV infusion, Q3W until disease progression, unacceptable toxicity, or withdrawal of consent, or for a maximum of 28.8 months.
- SCCHN: Part III Cohort K (QW/Q2W): CPI-naïve participants with SCCHN, received simlukafusp alfa, 10 mg, IV infusion, QW for the first 4 weeks, and Q2W until disease progression, unacceptable toxicity, or withdrawal of consent, or for a maximum of 24.3 months. Participants also received atezolizumab, 840 mg, IV infusion, Q2W in combination with simlukafusp alfa until disease progression, unacceptable toxicity, or withdrawal of consent, or for a maximum of 24.3 months.
- ESCC: Part III Cohort M (QW/Q2W): Participants with ESCC, received simlukafusp alfa, 10 mg, IV infusion, QW for the first 4 weeks, and Q2W until disease progression, unacceptable toxicity, or withdrawal of consent, or for a maximum of 4.1 months. Participants also received atezolizumab, 840 mg, IV infusion, Q2W in combination with simlukafusp alfa until disease progression, unacceptable toxicity, or withdrawal of consent, or for a maximum of 4.1 months.
- CSCC: Part III Cohort N (QW/Q2W): Participants with CSCC, received simlukafusp alfa, 10 mg, IV infusion, QW for the first 4 weeks, and Q2W until disease progression, unacceptable toxicity, or withdrawal of consent, or for a maximum of 0.68 months. Participants also received atezolizumab, 840 mg, IV infusion, Q2W in combination with simlukafusp alfa until disease progression, unacceptable toxicity, or withdrawal of consent, or for a maximum of 0.68 months.
Period: Overall Study
Arm/Group | NSCLC: Part I Cohort A (QW/Q2W) | NSCLC: Part I Cohort B (QW/Q2W) | NSCLC: Part I Cohort D, Arm 1 (QW/Q2W) | NSCLC: Part I Cohort D, Arm 2 (Q3W) | NSCLC: Part I Cohort D, Arm 3 (Q3W) | NSCLC: Part I Cohort F (Q3W) | NSCLC: Part II Cohort E, Arm 1 (QW/Q2W) | NSCLC: Part II Cohort E, Arm 2 (Q3W) | SCCHN: Part III Cohort G (Q3W) | SCCHN: Part III Cohort H (Q3W) | ESCC: Part III Cohort I (Q3W) | CSCC: Part III Cohort J (Q3W) | SCCHN: Part III Cohort K (QW/Q2W) | ESCC: Part III Cohort M (QW/Q2W) | CSCC: Part III Cohort N (QW/Q2W)
Started | 26 | 32 | 3 | 5 | 2 | 22 | 3 | 2 | 23 | 30 | 33 | 47 | 25 | 2 | 1
Response Evaluable Population (Response evaluable population included all participants in the safety population who received at least one dose of simlukafusp alfa/atezolizumab and who had at least one baseline and one on-study tumor assessment.) | 26 | 32 | 3 | 5 | 0 | 21 | 3 | 2 | 22 | 28 | 32 | 44 | 25 | 2 | 1
Completed | 4 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 6 | 0 | 0 | 0
Not Completed | 22 | 31 | 3 | 5 | 2 | 21 | 3 | 2 | 22 | 30 | 31 | 41 | 25 | 2 | 1
Not completed — Death | 12 | 21 | 2 | 5 | 1 | 12 | 1 | 1 | 12 | 20 | 21 | 21 | 14 | 2 | 1
Not completed — Lost to Follow-up | 1 | 3 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0
Not completed — Reason not specified | 3 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 1 | 2 | 6 | 1 | 0 | 0
Not completed — Progressive Disease | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 1 | 0 | 0
Not completed — Site Terminated by Sponsor | 5 | 5 | 0 | 0 | 1 | 3 | 0 | 1 | 4 | 5 | 3 | 11 | 6 | 0 | 0
Not completed — Symptomatic Deterioration | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 3 | 2 | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least one dose of study treatment, whether or not prematurely withdrawn from the study.
Groups:
- NSCLC: Part I Cohort A (QW/Q2W): CPI-naïve participants with NSCLC, received simlukafusp alfa, 10 mg, IV infusion, QW for the first 4 weeks, and Q2W until disease progression, unacceptable toxicity, or withdrawal of consent, or for a maximum of 38 months. Participants also received atezolizumab, 840 mg, IV infusion, Q2W in combination with simlukafusp alfa until disease progression, unacceptable toxicity, or withdrawal of consent, or for a maximum of 38 months.
- NSCLC: Part I Cohort D, Arm 2 (Q3W): CPI-experienced participants with NSCLC previously treated with platinum-containing regimen and docetaxel received simlukafusp alfa, 10 mg, IV infusion Q3W in combination with atezolizumab, 1200 mg, IV infusion, Q3W until disease progression, unacceptable toxicity, or withdrawal of consent, or for a maximum of 5.4 months.
- NSCLC: Part II Cohort E, Arm 1 (QW/Q2W): NSCLC participants without prior treatment for metastatic disease and with high PD-L1 expression levels, received simlukafusp alfa, 10 mg, IV infusion, QW for the first 4 weeks, and Q2W until disease progression, unacceptable toxicity, or withdrawal of consent, or for a maximum of 31.3 months. Participants also received atezolizumab, 840 mg, IV infusion, Q2W in combination with simlukafusp alfa until disease progression, unacceptable toxicity, or withdrawal of consent, or for a maximum of 31.3 months.
- Total: Total of all reporting groups
Arm/Group | NSCLC: Part I Cohort A (QW/Q2W) | NSCLC: Part I Cohort B (QW/Q2W) | NSCLC: Part I Cohort D, Arm 1 (QW/Q2W) | NSCLC: Part I Cohort D, Arm 2 (Q3W) | NSCLC: Part I Cohort D, Arm 3 (Q3W) | NSCLC: Part I Cohort F (Q3W) | NSCLC: Part II Cohort E, Arm 1 (QW/Q2W) | NSCLC: Part II Cohort E, Arm 2 (Q3W) | SCCHN: Part III Cohort G (Q3W) | SCCHN: Part III Cohort H (Q3W) | ESCC: Part III Cohort I (Q3W) | CSCC: Part III Cohort J (Q3W) | SCCHN: Part III Cohort K (QW/Q2W) | ESCC: Part III Cohort M (QW/Q2W) | CSCC: Part III Cohort N (QW/Q2W) | Total
Number analyzed (Participants) | 26 | 32 | 3 | 5 | 2 | 22 | 3 | 2 | 23 | 30 | 33 | 47 | 25 | 2 | 1 | 256
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.0 (10.5) | 59.8 (9.9) | 63.7 (3.8) | 65.6 (4.3) | 63.5 (4.9) | 57.4 (8.9) | 56.7 (0.6) | 68.0 (2.8) | 55.7 (12.8) | 58.8 (8.2) | 63.1 (9.6) | 51.3 (11.2) | 55.8 (11.7) | 67.0 (15.6) | 49.0 (NA) — Since only 1 participant was analyzed, the standard deviation (SD) could not be calculated. | 57.6 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 1 | 0 | 1 | 11 | 1 | 0 | 5 | 7 | 10 | 47 | 6 | 0 | 1 | 110
  Male | 16 | 22 | 2 | 5 | 1 | 11 | 2 | 2 | 18 | 23 | 23 | 0 | 19 | 2 | 0 | 146
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 9 | 5 | 0 | 0 | 0 | 5 | 1 | 0 | 3 | 5 | 6 | 0 | 5 | 1 | 0 | 40
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 4
  Black or African American | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
  White | 15 | 26 | 3 | 5 | 2 | 17 | 2 | 2 | 19 | 16 | 22 | 33 | 18 | 0 | 1 | 181
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 5 | 13 | 2 | 1 | 0 | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3
  Not Hispanic or Latino | 23 | 28 | 3 | 4 | 2 | 20 | 3 | 2 | 22 | 21 | 27 | 33 | 23 | 1 | 1 | 213
  Not Stated | 1 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 7 | 4 | 9 | 2 | 1 | 0 | 29
  Unknown | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 5 | 0 | 0 | 0 | 11

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Objective Response Rate (ORR) According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Description: ORR was defined as the percentage of participants with observed tumor response of complete response (CR), or partial response (PR) determined according to RECIST version 1.1. CR was defined as the disappearance of all target lesions with reduction in target/non-target pathological lymph nodes to <10 millimeters (mm). PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. The percentages of participants are rounded off to the nearest single decimal point.
Time Frame: Baseline up to disease progression or study treatment discontinuation (up to 38 months)
Population: Response evaluable population included all participants in the safety population who received at least one dose of simlukafusp alfa/atezolizumab and who had at least one baseline and one on-study tumor assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | NSCLC: Part I Cohort A (QW/Q2W) | NSCLC: Part I Cohort B (QW/Q2W) | NSCLC: Part I Cohort D, Arm 1 (QW/Q2W) | NSCLC: Part I Cohort D, Arm 2 (Q3W) | NSCLC: Part I Cohort D, Arm 3 (Q3W) | NSCLC: Part I Cohort F (Q3W) | NSCLC: Part II Cohort E, Arm 1 (QW/Q2W) | NSCLC: Part II Cohort E, Arm 2 (Q3W) | SCCHN: Part III Cohort G (Q3W) | SCCHN: Part III Cohort H (Q3W) | ESCC: Part III Cohort I (Q3W) | CSCC: Part III Cohort J (Q3W) | SCCHN: Part III Cohort K (QW/Q2W) | ESCC: Part III Cohort M (QW/Q2W) | CSCC: Part III Cohort N (QW/Q2W)
Number analyzed (Participants) | 26 | 32 | 3 | 5 | 0 | 21 | 3 | 2 | 22 | 28 | 32 | 44 | 25 | 2 | 1
percentage of participants | 19.2 [8.51 to 37.88] | 6.3 [1.73 to 20.15] | 0 [0.00 to 56.15] | 0 [0.00 to 43.45] |  | 4.8 [0.85 to 22.67] | 66.7 [20.77 to 93.85] | 50.0 [9.45 to 90.55] | 18.2 [7.31 to 38.52] | 3.6 [0.63 to 17.71] | 21.9 [11.02 to 38.75] | 27.3 [16.35 to 41.85] | 4.0 [0.71 to 19.54] | 0 [0.00 to 65.76] | 0 [0.00 to 79.35]

2. Secondary Outcome: Percentage of Participants With Disease Control Rate (DCR) Determined According to RECIST Version 1.1
Description: DCR was defined as the percentage of participants with observed tumor response of CR, PR or stable disease (SD) determined according to RECIST version 1.1. CR was defined as the disappearance of all target lesions with reduction in target/non-target pathological lymph nodes to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD). PD is at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study including baseline (nadir). The percentages of participants are rounded off to the nearest single decimal point.
Time Frame: Baseline up to disease progression or study treatment discontinuation (up to 38 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | NSCLC: Part I Cohort A (QW/Q2W) | NSCLC: Part I Cohort B (QW/Q2W) | NSCLC: Part I Cohort D, Arm 1 (QW/Q2W) | NSCLC: Part I Cohort D, Arm 2 (Q3W) | NSCLC: Part I Cohort D, Arm 3 (Q3W) | NSCLC: Part I Cohort F (Q3W) | NSCLC: Part II Cohort E, Arm 1 (QW/Q2W) | NSCLC: Part II Cohort E, Arm 2 (Q3W) | SCCHN: Part III Cohort G (Q3W) | SCCHN: Part III Cohort H (Q3W) | ESCC: Part III Cohort I (Q3W) | CSCC: Part III Cohort J (Q3W) | SCCHN: Part III Cohort K (QW/Q2W) | ESCC: Part III Cohort M (QW/Q2W) | CSCC: Part III Cohort N (QW/Q2W)
Number analyzed (Participants) | 26 | 32 | 3 | 5 | 0 | 21 | 3 | 2 | 22 | 28 | 32 | 44 | 25 | 2 | 1
percentage of participants | 53.8 [35.46 to 71.24] | 62.5 [45.25 to 77.07] | 0 [0.00 to 56.15] | 20.0 [3.62 to 62.45] |  | 57.1 [36.55 to 75.53] | 66.7 [20.77 to 93.85] | 50.0 [9.45 to 90.55] | 50.0 [30.72 to 69.28] | 14.3 [5.70 to 31.49] | 43.8 [28.17 to 60.67] | 68.2 [53.44 to 80.00] | 36.0 [20.25 to 55.48] | 50.0 [9.45 to 90.55] | 0 [0.00 to 79.35]

3. Secondary Outcome: Duration of Response (DoR) According to RECIST Version 1.1
Description: DoR was determined for participants who had a best overall response of CR or PR. CR was defined as the disappearance of all target lesions with a reduction in target/non-target pathological lymph nodes to < 10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. DoR was defined as the time from first occurrence of a documented objective response until the time of documented disease progression or death from any cause during treatment, whichever occurs first. Participants that did not have documented progressive disease or death during the study were censored at the day of the last tumor assessment.
Time Frame: From first occurrence of documented CR or PR up to disease progression or study treatment discontinuation (assessed every 8 weeks after study treatment start for the first year, and every 12 weeks thereafter, up to 38 months)
Population: Data was not collected for this outcome measure due to premature termination of the study by the sponsor.
Arm/Group | NSCLC: Part I Cohort A (QW/Q2W) | NSCLC: Part I Cohort B (QW/Q2W) | NSCLC: Part I Cohort D, Arm 1 (QW/Q2W) | NSCLC: Part I Cohort D, Arm 2 (Q3W) | NSCLC: Part I Cohort D, Arm 3 (Q3W) | NSCLC: Part I Cohort F (Q3W) | NSCLC: Part II Cohort E, Arm 1 (QW/Q2W) | NSCLC: Part II Cohort E, Arm 2 (Q3W) | SCCHN: Part III Cohort G (Q3W) | SCCHN: Part III Cohort H (Q3W) | ESCC: Part III Cohort I (Q3W) | CSCC: Part III Cohort J (Q3W) | SCCHN: Part III Cohort K (QW/Q2W) | ESCC: Part III Cohort M (QW/Q2W) | CSCC: Part III Cohort N (QW/Q2W)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Progression-Free Survival (PFS) According to RECIST Version 1.1
Description: PFS was defined as the time from study treatment initiation (Cycle 1 Day 1 [1 cycle=14 days for QW/Q2W cohorts; 1 cycle=21 days for Q3W cohorts]) to the first occurrence of documented disease progression (based on Investigator's assessment) or death from any cause during treatment, whichever occurs first. Participants that did not have documented progressive disease or death during the study were censored at the day of the last tumor assessment.
Time Frame: Study treatment initiation up to disease progression or study treatment discontinuation (up to 38 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | NSCLC: Part I Cohort A (QW/Q2W) | NSCLC: Part I Cohort B (QW/Q2W) | NSCLC: Part I Cohort D, Arm 1 (QW/Q2W) | NSCLC: Part I Cohort D, Arm 2 (Q3W) | NSCLC: Part I Cohort D, Arm 3 (Q3W) | NSCLC: Part I Cohort F (Q3W) | NSCLC: Part II Cohort E, Arm 1 (QW/Q2W) | NSCLC: Part II Cohort E, Arm 2 (Q3W) | SCCHN: Part III Cohort G (Q3W) | SCCHN: Part III Cohort H (Q3W) | ESCC: Part III Cohort I (Q3W) | CSCC: Part III Cohort J (Q3W) | SCCHN: Part III Cohort K (QW/Q2W) | ESCC: Part III Cohort M (QW/Q2W) | CSCC: Part III Cohort N (QW/Q2W)
Number analyzed (Participants) | 26 | 32 | 3 | 5 | 0 | 21 | 3 | 2 | 22 | 28 | 32 | 44 | 25 | 2 | 1
months | 3.5 [1.7 to 7.4] | 3.7 [3.1 to 5.2] | 2.0 [1.7 to NA] — Upper limit of 95% confidence interval (CI) could not be calculated due to low number of participants with events. | 2.0 [1.9 to NA] — Upper limit of 95% CI could not be calculated due to low number of participants with events. |  | 3.5 [1.9 to 5.5] | NA [2.6 to NA] — Median and Upper limit of 95% CI could not be calculated due to low number of participants with events. | 10.5 [1.9 to NA] — Upper limit of 95% CI could not be calculated due to low number of participants with events. | 2.5 [1.8 to 5.6] | 1.9 [1.8 to 1.9] | 1.9 [1.8 to 3.7] | 3.7 [3.3 to 9.0] | 1.9 [1.6 to 3.2] | 2.6 [1.6 to NA] — Upper limit of 95% CI could not be calculated due to low number of participants with events. | 1.9 [NA to NA] — Upper and lower limit of 95% CI could not be calculated as only one participant with events was evaluated.

5. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the first dose of study treatment to the time of death from any cause on study. Participants who were still alive at the time of analysis were censored at the last date known alive.
Time Frame: From first dose of study treatment up to death due to any cause (up to approximately 47 months)
Population: Response evaluable population included all participants in the safety population who received at least one dose of simlukafusp alfa/atezolizumab and who had at least one baseline and one on-study tumor assessment. Due to early termination of the study, matured median for OS could not be achieved, hence as planned and pre-specified in the protocol, the data for OS was not analyzed and not reported.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | NSCLC: Part I Cohort A (QW/Q2W) | NSCLC: Part I Cohort B (QW/Q2W) | NSCLC: Part I Cohort D, Arm 1 (QW/Q2W) | NSCLC: Part I Cohort D, Arm 2 (Q3W) | NSCLC: Part I Cohort D, Arm 3 (Q3W) | NSCLC: Part I Cohort F (Q3W) | NSCLC: Part II Cohort E, Arm 1 (QW/Q2W) | NSCLC: Part II Cohort E, Arm 2 (Q3W) | SCCHN: Part III Cohort G (Q3W) | SCCHN: Part III Cohort H (Q3W) | ESCC: Part III Cohort I (Q3W) | CSCC: Part III Cohort J (Q3W) | SCCHN: Part III Cohort K (QW/Q2W) | ESCC: Part III Cohort M (QW/Q2W) | CSCC: Part III Cohort N (QW/Q2W)
Number analyzed (Participants) | 26 | 32 | 3 | 5 | 0 | 21 | 3 | 2 | 22 | 28 | 32 | 44 | 25 | 2 | 1
months | NA [NA to NA] — Due to early termination of the study, matured median for OS could not be achieved, hence as planned and pre-specified in the protocol, the data for OS was not analyzed and not reported. | NA [NA to NA] — Due to early termination of the study, matured median for OS could not be achieved, hence as planned and pre-specified in the protocol, the data for OS was not analyzed and not reported. | NA [NA to NA] — Due to early termination of the study, matured median for OS could not be achieved, hence as planned and pre-specified in the protocol, the data for OS was not analyzed and not reported. | NA [NA to NA] — Due to early termination of the study, matured median for OS could not be achieved, hence as planned and pre-specified in the protocol, the data for OS was not analyzed and not reported. |  | NA [NA to NA] — Due to early termination of the study, matured median for OS could not be achieved, hence as planned and pre-specified in the protocol, the data for OS was not analyzed and not reported. | NA [NA to NA] — Due to early termination of the study, matured median for OS could not be achieved, hence as planned and pre-specified in the protocol, the data for OS was not analyzed and not reported. | NA [NA to NA] — Due to early termination of the study, matured median for OS could not be achieved, hence as planned and pre-specified in the protocol, the data for OS was not analyzed and not reported. | NA [NA to NA] — Due to early termination of the study, matured median for OS could not be achieved, hence as planned and pre-specified in the protocol, the data for OS was not analyzed and not reported. | NA [NA to NA] — Due to early termination of the study, matured median for OS could not be achieved, hence as planned and pre-specified in the protocol, the data for OS was not analyzed and not reported. | NA [NA to NA] — Due to early termination of the study, matured median for OS could not be achieved, hence as planned and pre-specified in the protocol, the data for OS was not analyzed and not reported. | NA [NA to NA] — Due to early termination of the study, matured median for OS could not be achieved, hence as planned and pre-specified in the protocol, the data for OS was not analyzed and not reported. | NA [NA to NA] — Due to early termination of the study, matured median for OS could not be achieved, hence as planned and pre-specified in the protocol, the data for OS was not analyzed and not reported. | NA [NA to NA] — Due to early termination of the study, matured median for OS could not be achieved, hence as planned and pre-specified in the protocol, the data for OS was not analyzed and not reported. | NA [NA to NA] — Due to early termination of the study, matured median for OS could not be achieved, hence as planned and pre-specified in the protocol, the data for OS was not analyzed and not reported.

6. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: Baseline up to end of the study (up to approximately 47 months)
Population: Safety Population included all participants who received at least one dose of study treatment, whether prematurely withdrawn from the study or not.
Measure: Number; unit: percentage of participants
Arm/Group | NSCLC: Part I Cohort A (QW/Q2W) | NSCLC: Part I Cohort B (QW/Q2W) | NSCLC: Part I Cohort D, Arm 1 (QW/Q2W) | NSCLC: Part I Cohort D, Arm 2 (Q3W) | NSCLC: Part I Cohort D, Arm 3 (Q3W) | NSCLC: Part I Cohort F (Q3W) | NSCLC: Part II Cohort E, Arm 1 (QW/Q2W) | NSCLC: Part II Cohort E, Arm 2 (Q3W) | SCCHN: Part III Cohort G (Q3W) | SCCHN: Part III Cohort H (Q3W) | ESCC: Part III Cohort I (Q3W) | CSCC: Part III Cohort J (Q3W) | SCCHN: Part III Cohort K (QW/Q2W) | ESCC: Part III Cohort M (QW/Q2W) | CSCC: Part III Cohort N (QW/Q2W)
Number analyzed (Participants) | 26 | 32 | 3 | 5 | 2 | 22 | 3 | 2 | 23 | 30 | 33 | 47 | 25 | 2 | 1
percentage of participants | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100

7. Secondary Outcome: Percentage of Participants by Programmed Death-Ligand 1 (PD-L1) Status According to Immunohistochemical Methods
Time Frame: Baseline
Population: Data was not collected for this outcome measure post-baseline as baseline data was not matured and sufficient to analyze PD-L1 impact.
Arm/Group | NSCLC: Part I Cohort A (QW/Q2W) | NSCLC: Part I Cohort B (QW/Q2W) | NSCLC: Part I Cohort D, Arm 1 (QW/Q2W) | NSCLC: Part I Cohort D, Arm 2 (Q3W) | NSCLC: Part I Cohort D, Arm 3 (Q3W) | NSCLC: Part I Cohort F (Q3W) | NSCLC: Part II Cohort E, Arm 1 (QW/Q2W) | NSCLC: Part II Cohort E, Arm 2 (Q3W) | SCCHN: Part III Cohort G (Q3W) | SCCHN: Part III Cohort H (Q3W) | ESCC: Part III Cohort I (Q3W) | CSCC: Part III Cohort J (Q3W) | SCCHN: Part III Cohort K (QW/Q2W) | ESCC: Part III Cohort M (QW/Q2W) | CSCC: Part III Cohort N (QW/Q2W)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Change From Baseline in Density of Cluster of Differentiation (CD) 8 Positive (CD8+) Cells According to Immunohistochemical Methods
Time Frame: Baseline up 2 months
Population: Data was not collected for this outcome measure post-baseline as baseline data was not matured and sufficient to be analyzed during analysis.
Arm/Group | NSCLC: Part I Cohort A (QW/Q2W) | NSCLC: Part I Cohort B (QW/Q2W) | NSCLC: Part I Cohort D, Arm 1 (QW/Q2W) | NSCLC: Part I Cohort D, Arm 2 (Q3W) | NSCLC: Part I Cohort D, Arm 3 (Q3W) | NSCLC: Part I Cohort F (Q3W) | NSCLC: Part II Cohort E, Arm 1 (QW/Q2W) | NSCLC: Part II Cohort E, Arm 2 (Q3W) | SCCHN: Part III Cohort G (Q3W) | SCCHN: Part III Cohort H (Q3W) | ESCC: Part III Cohort I (Q3W) | CSCC: Part III Cohort J (Q3W) | SCCHN: Part III Cohort K (QW/Q2W) | ESCC: Part III Cohort M (QW/Q2W) | CSCC: Part III Cohort N (QW/Q2W)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Change From Baseline in Density of Cluster of Differentiation 3 Negative (CD3-) Perforin Positive Cells According to Immunohistochemical Methods
Time Frame: Baseline up to 2 months
Population: as for outcome 8
Arm/Group | NSCLC: Part I Cohort A (QW/Q2W) | NSCLC: Part I Cohort B (QW/Q2W) | NSCLC: Part I Cohort D, Arm 1 (QW/Q2W) | NSCLC: Part I Cohort D, Arm 2 (Q3W) | NSCLC: Part I Cohort D, Arm 3 (Q3W) | NSCLC: Part I Cohort F (Q3W) | NSCLC: Part II Cohort E, Arm 1 (QW/Q2W) | NSCLC: Part II Cohort E, Arm 2 (Q3W) | SCCHN: Part III Cohort G (Q3W) | SCCHN: Part III Cohort H (Q3W) | ESCC: Part III Cohort I (Q3W) | CSCC: Part III Cohort J (Q3W) | SCCHN: Part III Cohort K (QW/Q2W) | ESCC: Part III Cohort M (QW/Q2W) | CSCC: Part III Cohort N (QW/Q2W)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Change From Baseline in Density of PD-L1 According to Immunohistochemical Methods
Time Frame: Baseline up to 2 months
Population: as for outcome 7
Arm/Group | NSCLC: Part I Cohort A (QW/Q2W) | NSCLC: Part I Cohort B (QW/Q2W) | NSCLC: Part I Cohort D, Arm 1 (QW/Q2W) | NSCLC: Part I Cohort D, Arm 2 (Q3W) | NSCLC: Part I Cohort D, Arm 3 (Q3W) | NSCLC: Part I Cohort F (Q3W) | NSCLC: Part II Cohort E, Arm 1 (QW/Q2W) | NSCLC: Part II Cohort E, Arm 2 (Q3W) | SCCHN: Part III Cohort G (Q3W) | SCCHN: Part III Cohort H (Q3W) | ESCC: Part III Cohort I (Q3W) | CSCC: Part III Cohort J (Q3W) | SCCHN: Part III Cohort K (QW/Q2W) | ESCC: Part III Cohort M (QW/Q2W) | CSCC: Part III Cohort N (QW/Q2W)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to end of the study (up to approximately 47 months)
Description: Safety-evaluable population included all participants who received at least one dose of study treatment, whether prematurely withdrawn from the study or not.
Arm/Group | NSCLC: Part I Cohort A (QW/Q2W) | NSCLC: Part I Cohort B (QW/Q2W) | NSCLC: Part I Cohort D, Arm 1 (QW/Q2W) | NSCLC: Part I Cohort D, Arm 2 (Q3W) | NSCLC: Part I Cohort D, Arm 3 (Q3W) | NSCLC: Part I Cohort F (Q3W) | NSCLC: Part II Cohort E, Arm 1 (QW/Q2W) | NSCLC: Part II Cohort E, Arm 2 (Q3W) | SCCHN: Part III Cohort G (Q3W) | SCCHN: Part III Cohort H (Q3W) | ESCC: Part III Cohort I (Q3W) | CSCC: Part III Cohort J (Q3W) | SCCHN: Part III Cohort K (QW/Q2W) | ESCC: Part III Cohort M (QW/Q2W) | CSCC: Part III Cohort N (QW/Q2W)
All-Cause Mortality (participants affected / at risk) | 12/26 | 21/32 | 3/3 | 5/5 | 1/2 | 12/22 | 1/3 | 1/2 | 14/23 | 20/30 | 21/33 | 21/47 | 14/25 | 2/2 | 1/1
Serious Adverse Events (participants affected / at risk) | 13/26 | 25/32 | 0/3 | 3/5 | 2/2 | 14/22 | 1/3 | 1/2 | 15/23 | 22/30 | 20/33 | 32/47 | 14/25 | 1/2 | 1/1
Other Adverse Events (participants affected / at risk) | 25/26 | 32/32 | 3/3 | 5/5 | 2/2 | 21/22 | 3/3 | 2/2 | 23/23 | 29/30 | 33/33 | 47/47 | 24/25 | 2/2 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NSCLC: Part I Cohort A (QW/Q2W) (N=26) | NSCLC: Part I Cohort B (QW/Q2W) (N=32) | NSCLC: Part I Cohort D, Arm 1 (QW/Q2W) (N=3) | NSCLC: Part I Cohort D, Arm 2 (Q3W) (N=5) | NSCLC: Part I Cohort D, Arm 3 (Q3W) (N=2) | NSCLC: Part I Cohort F (Q3W) (N=22) | NSCLC: Part II Cohort E, Arm 1 (QW/Q2W) (N=3) | NSCLC: Part II Cohort E, Arm 2 (Q3W) (N=2) | SCCHN: Part III Cohort G (Q3W) (N=23) | SCCHN: Part III Cohort H (Q3W) (N=30) | ESCC: Part III Cohort I (Q3W) (N=33) | CSCC: Part III Cohort J (Q3W) (N=47) | SCCHN: Part III Cohort K (QW/Q2W) (N=25) | ESCC: Part III Cohort M (QW/Q2W) (N=2) | CSCC: Part III Cohort N (QW/Q2W) (N=1)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 2 (3) | 2 (2) | 0 (0) | 0 (0)
LYMPHOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 1 (2) | 0 (0) | 2 (4) | 1 (1) | 0 (0) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MYOCARDITIS (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PERICARDIAL EFFUSION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TRACHEO-OESOPHAGEAL FISTULA (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ADDISON'S DISEASE (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
IMMUNE-MEDIATED HYPOPHYSITIS (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COLITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTRIC HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
IMMUNE-MEDIATED ENTEROCOLITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LARGE INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MOUTH HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OESOPHAGEAL FISTULA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OESOPHAGEAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OESOPHAGEAL STENOSIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PANCREATITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PROCTALGIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CHILLS (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FACIAL PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GENERALISED OEDEMA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFLAMMATION (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFLUENZA LIKE ILLNESS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
MALAISE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MEDICAL DEVICE SITE HAEMORRHAGE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
OEDEMA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PAIN (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PERFORMANCE STATUS DECREASED (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (2) | 4 (6) | 1 (1) | 0 (0) | 0 (0)
BILE DUCT STENOSIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
BILIARY OBSTRUCTION (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DRUG-INDUCED LIVER INJURY (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEPATITIS (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEPATOTOXICITY (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANAPHYLACTIC REACTION (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANAPHYLACTIC SHOCK (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SYSTEMIC IMMUNE ACTIVATION (Immune system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL WALL ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
APPENDICITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ARTHRITIS BACTERIAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ASPERGILLUS INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BACTERAEMIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
BACTERIAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BRONCHITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CORNEAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
DEVICE RELATED INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
ENCEPHALITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ESCHERICHIA INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LYMPH GLAND INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PELVIC INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PERITONEAL ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PLEURAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
PNEUMONIA BACTERIAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA NECROTISING (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PULMONARY SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SEPTIC SHOCK (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SKIN INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
VASCULAR DEVICE INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INCORRECT DOSE ADMINISTERED (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 0 (0) | 3 (17) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 3 (3) | 1 (1) | 7 (12) | 4 (9) | 0 (0) | 0 (0)
MEDICATION ERROR (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SKIN LACERATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UROSTOMY COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VASCULAR ACCESS COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD BILIRUBIN INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD CREATININE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
EJECTION FRACTION DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HEPATIC ENZYME INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LIVER FUNCTION TEST ABNORMAL (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LIVER FUNCTION TEST INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LYMPHOCYTE COUNT DECREASED (Investigations) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OXYGEN SATURATION DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PLATELET COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
TRANSAMINASES INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MALNUTRITION (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TYPE 1 DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MALIGNANT NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
TUMOUR HAEMORRHAGE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TUMOUR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
AGNOSIA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
APHASIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CEREBRAL ISCHAEMIA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
EPILEPSY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEURALGIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
POLYNEUROPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SYNCOPE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
VOCAL CORD PARALYSIS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DEVICE DISLOCATION (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CONFUSIONAL STATE (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYDRONEPHROSIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
NEPHRITIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PYELOCALIECTASIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RENAL FAILURE (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FEMALE GENITAL TRACT FISTULA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LARYNGEAL HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PHARYNGEAL HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
STEVENS-JOHNSON SYNDROME (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MEDICAL DEVICE REMOVAL (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CAPILLARY LEAK SYNDROME (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
EMBOLISM (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOTENSION (Vascular disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VASCULITIS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NSCLC: Part I Cohort A (QW/Q2W) (N=26) | NSCLC: Part I Cohort B (QW/Q2W) (N=32) | NSCLC: Part I Cohort D, Arm 1 (QW/Q2W) (N=3) | NSCLC: Part I Cohort D, Arm 2 (Q3W) (N=5) | NSCLC: Part I Cohort D, Arm 3 (Q3W) (N=2) | NSCLC: Part I Cohort F (Q3W) (N=22) | NSCLC: Part II Cohort E, Arm 1 (QW/Q2W) (N=3) | NSCLC: Part II Cohort E, Arm 2 (Q3W) (N=2) | SCCHN: Part III Cohort G (Q3W) (N=23) | SCCHN: Part III Cohort H (Q3W) (N=30) | ESCC: Part III Cohort I (Q3W) (N=33) | CSCC: Part III Cohort J (Q3W) (N=47) | SCCHN: Part III Cohort K (QW/Q2W) (N=25) | ESCC: Part III Cohort M (QW/Q2W) (N=2) | CSCC: Part III Cohort N (QW/Q2W) (N=1)
ANAEMIA (Blood and lymphatic system disorders) | 3 (3) | 11 (18) | 0 (0) | 1 (3) | 0 (0) | 5 (7) | 0 (0) | 0 (0) | 15 (29) | 9 (13) | 7 (8) | 23 (40) | 11 (29) | 0 (0) | 0 (0)
COAGULOPATHY (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
LEUKOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 3 (11) | 2 (2) | 0 (0) | 0 (0)
LYMPHOCYTOSIS (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LYMPHOPENIA (Blood and lymphatic system disorders) | 0 (0) | 4 (7) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (8) | 0 (0) | 4 (15) | 3 (7) | 3 (17) | 6 (17) | 4 (25) | 0 (0) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 3 (5) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 6 (12) | 3 (4) | 0 (0) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (4) | 6 (14) | 2 (2) | 0 (0) | 0 (0)
CARDIAC FAILURE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GLUCOCORTICOID DEFICIENCY (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERTHYROIDISM (Endocrine disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
HYPOTHYROIDISM (Endocrine disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 4 (4) | 1 (1) | 7 (7) | 3 (4) | 5 (5) | 0 (0) | 0 (0)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 10 (12) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 5 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 5 (6) | 4 (5) | 6 (7) | 6 (9) | 0 (0) | 2 (2) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 9 (17) | 9 (10) | 2 (2) | 0 (0) | 0 (0) | 3 (4) | 1 (2) | 0 (0) | 3 (3) | 5 (6) | 7 (7) | 17 (29) | 4 (4) | 1 (2) | 0 (0)
DRY MOUTH (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (12) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 11 (22) | 10 (11) | 1 (2) | 0 (0) | 0 (0) | 8 (11) | 2 (2) | 0 (0) | 6 (14) | 7 (11) | 13 (49) | 19 (46) | 11 (44) | 0 (0) | 1 (1)
OESOPHAGEAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
STOMATITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
TOOTHACHE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 10 (24) | 7 (10) | 1 (3) | 1 (1) | 0 (0) | 11 (16) | 0 (0) | 0 (0) | 5 (19) | 5 (6) | 3 (4) | 18 (45) | 1 (1) | 0 (0) | 1 (2)
ASTHENIA (General disorders) | 6 (9) | 7 (8) | 2 (3) | 2 (2) | 1 (1) | 7 (8) | 1 (2) | 0 (0) | 9 (10) | 12 (12) | 8 (8) | 23 (28) | 4 (4) | 0 (0) | 0 (0)
CHEST PAIN (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
CHILLS (General disorders) | 12 (23) | 12 (23) | 1 (1) | 2 (4) | 0 (0) | 9 (15) | 1 (3) | 0 (0) | 6 (8) | 10 (10) | 12 (25) | 12 (18) | 9 (49) | 2 (7) | 1 (3)
FATIGUE (General disorders) | 14 (25) | 15 (21) | 0 (0) | 1 (1) | 0 (0) | 3 (6) | 1 (4) | 1 (1) | 6 (9) | 5 (6) | 8 (11) | 9 (12) | 11 (19) | 0 (0) | 1 (1)
HYPERTHERMIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFLUENZA LIKE ILLNESS (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (23) | 0 (0) | 0 (0) | 0 (0)
MALAISE (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
MUCOSAL INFLAMMATION (General disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 2 (2) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
OEDEMA (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 6 (6) | 4 (7) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (2) | 7 (9) | 0 (0) | 0 (0) | 0 (0)
PAIN (General disorders) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 20 (197) | 29 (91) | 3 (11) | 5 (11) | 1 (3) | 15 (47) | 2 (7) | 1 (3) | 18 (76) | 22 (60) | 26 (116) | 35 (134) | 21 (110) | 2 (13) | 1 (4)
XEROSIS (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEPATOTOXICITY (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 0 (0)
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 1 (2) | 2 (8) | 3 (4) | 0 (0) | 0 (0)
BACTERAEMIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BRONCHITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CELLULITIS (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CONJUNCTIVITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ORAL CANDIDIASIS (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RHINITIS (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 (5) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (5) | 14 (19) | 1 (2) | 0 (0) | 0 (0)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 4 (11) | 7 (16) | 0 (0) | 2 (2) | 0 (0) | 2 (4) | 1 (1) | 0 (0) | 2 (13) | 1 (3) | 5 (23) | 7 (16) | 5 (24) | 0 (0) | 0 (0)
TOOTH FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 9 (24) | 9 (12) | 0 (0) | 1 (1) | 0 (0) | 3 (7) | 1 (1) | 1 (1) | 12 (21) | 6 (7) | 14 (27) | 21 (49) | 9 (13) | 0 (0) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 12 (27) | 8 (13) | 0 (0) | 1 (1) | 0 (0) | 5 (9) | 1 (1) | 1 (1) | 16 (37) | 6 (9) | 14 (25) | 22 (56) | 11 (21) | 1 (1) | 0 (0)
BILIRUBIN CONJUGATED INCREASED (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 4 (9) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 7 (15) | 4 (5) | 5 (7) | 11 (18) | 8 (15) | 0 (0) | 0 (0)
BLOOD BILIRUBIN INCREASED (Investigations) | 6 (15) | 6 (11) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (10) | 0 (0) | 5 (10) | 2 (4) | 6 (7) | 12 (14) | 6 (6) | 0 (0) | 0 (0)
BLOOD CHOLESTEROL INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD CREATININE INCREASED (Investigations) | 3 (6) | 4 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (8) | 1 (3) | 1 (1) | 6 (7) | 3 (3) | 0 (0) | 0 (0)
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 2 (5) | 6 (8) | 4 (6) | 0 (0) | 0 (0)
BLOOD URIC ACID INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
C-REACTIVE PROTEIN INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
EOSINOPHIL COUNT INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 5 (5) | 4 (9) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (4) | 0 (0) | 12 (28) | 9 (9) | 5 (7) | 16 (25) | 12 (17) | 0 (0) | 0 (0)
HEPATIC ENZYME INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
LIPASE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LIVER FUNCTION TEST ABNORMAL (Investigations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
LYMPHOCYTE COUNT DECREASED (Investigations) | 2 (8) | 1 (6) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (10) | 0 (0) | 3 (9) | 5 (9) | 2 (16) | 0 (0) | 0 (0)
NEUTROPHIL COUNT DECREASED (Investigations) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 0 (0)
PLATELET COUNT DECREASED (Investigations) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 6 (24) | 2 (2) | 2 (6) | 5 (7) | 4 (8) | 0 (0) | 0 (0)
TRANSAMINASES INCREASED (Investigations) | 3 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
WEIGHT DECREASED (Investigations) | 6 (7) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 2 (2) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
WEIGHT INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (10) | 0 (0) | 0 (0) | 1 (2) | 2 (9) | 0 (0) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 7 (11) | 12 (16) | 2 (3) | 1 (1) | 1 (1) | 6 (6) | 2 (3) | 0 (0) | 4 (5) | 11 (11) | 6 (8) | 12 (15) | 3 (3) | 0 (0) | 0 (0)
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (8) | 2 (4) | 3 (3) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
HYPERNATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERURICAEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 5 (9) | 2 (2) | 1 (5) | 6 (10) | 2 (3) | 0 (0) | 0 (0)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (6) | 1 (1) | 0 (0) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 4 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 3 (5) | 2 (2) | 9 (11) | 2 (2) | 0 (0) | 0 (0)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 3 (14) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 4 (5) | 4 (6) | 2 (3) | 8 (13) | 2 (2) | 0 (0) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 8 (13) | 2 (2) | 2 (4) | 2 (4) | 4 (7) | 0 (0) | 0 (0)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 5 (12) | 4 (15) | 0 (0) | 1 (4) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 5 (11) | 5 (8) | 4 (13) | 9 (9) | 5 (7) | 0 (0) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 5 (6) | 7 (9) | 3 (7) | 0 (0) | 0 (0)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 7 (8) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 9 (10) | 0 (0) | 0 (0) | 1 (1)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 0 (0)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (8) | 0 (0) | 4 (4) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 7 (7) | 0 (0) | 0 (0) | 0 (0)
TUMOUR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 3 (5) | 1 (1) | 0 (0) | 0 (0)
DYSGEUSIA (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 4 (8) | 4 (6) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 2 (3) | 0 (0) | 2 (3) | 1 (1) | 7 (13) | 8 (9) | 4 (10) | 1 (1) | 1 (1)
HYPOAESTHESIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
NEUROTOXICITY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PRESYNCOPE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANXIETY (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
CONFUSIONAL STATE (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INSOMNIA (Psychiatric disorders) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 3 (5) | 8 (9) | 1 (1) | 0 (0) | 0 (0)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
PROTEINURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (5) | 0 (0) | 0 (0)
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (5) | 1 (7) | 0 (0) | 0 (0) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 8 (11) | 2 (2) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 4 (5) | 6 (6) | 2 (2) | 0 (0) | 0 (0)
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 7 (10) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 4 (5) | 6 (8) | 2 (3) | 0 (0) | 0 (0)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
DERMATITIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DRY SKIN (Skin and subcutaneous tissue disorders) | 2 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 3 (7) | 1 (1) | 1 (1) | 0 (0)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 3 (3) | 2 (7) | 0 (0) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 6 (11) | 6 (8) | 2 (2) | 2 (2) | 0 (0) | 7 (8) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 4 (7) | 8 (9) | 7 (9) | 1 (2) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 13 (26) | 5 (5) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 2 (6) | 0 (0) | 7 (12) | 1 (1) | 4 (7) | 9 (15) | 4 (5) | 1 (2) | 0 (0)
RASH MACULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 0 (0) | 0 (0)
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URTICARIA (Skin and subcutaneous tissue disorders) | 2 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
CAPILLARY LEAK SYNDROME (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HOT FLUSH (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPERTENSION (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (2) | 2 (4) | 1 (1) | 0 (0)
HYPOTENSION (Vascular disorders) | 2 (2) | 11 (14) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 0 (0) | 0 (0) | 4 (5) | 8 (11) | 2 (3) | 6 (8) | 3 (3) | 0 (0) | 0 (0)
THROMBOSIS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-21): https://cdn.clinicaltrials.gov/large-docs/21/NCT03386721/Prot_SAP_000.pdf